CLINICAL TRIAL: NCT05939141
Title: A Prospective, Open-label, Multicentric Extension Study to Assess the Long-term Safety of the Genio® System in Study Subjects Who Have Been Implanted With the Genio® Implantable Stimulator (IS) for the Treatment of OSA in Adult Patients.
Brief Title: An Extension Study to Assess the Long-term Safety of the Genio® System
Acronym: OLE
Status: Not yet recruiting | Type: Observational
Sponsor: Nyxoah S.A. (Industry)
Collaborators: Nyxoah Pty. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-OLE2023
Record Dates: First submitted 2023-06-16; First posted 2023-07-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: OSA HGNS Hypoglossal Nerve Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OLE Subjects: adult OSA patients with and without complete concentric collapse of the soft palate who have successfully been implanted with the Genio IS in a Nyxoah sponsored Clinical Investigation and having the device in-situ at the time of enrollment (with therapy activated or de-activated).
  Interventions: Device: Genio System

INTERVENTIONS:
Device: Genio System — All participants have previously been implanted with a Genio® system implantable stimulator. This research is observational in nature (long term safety follow-up) and participants will not be exposed to additional procedures.
  The Genio System comprises of a bilateral Implantable Stimulator (IS), which is implanted via a minimally invasive surgery procedure and positioned over the genioglossus muscle with its electrodes positioned over both the left and right hypoglossal nerve branches. Stimulation of the hypoglossal nerve causes the tongue muscles to contract with the intention to maintain an open airway. The Implantable Stimulator receives energy pulses transmitted via the DP placed under the patient's chin and connected to the Activation Chip (AC), which contains the patient's stimulation parameters and contain a battery that provides energy.

SUMMARY:
The objective of this study is to assess the long-term safety of the Genio® system in adult OSA patients with and without complete concentric collapse of the soft palate who have successfully been implanted with the Genio IS in a Nyxoah sponsored Clinical Investigation.

(Serious) Adverse Device Effects and Device Deficiencies in subjects previously implanted with a Nyxoah Genio implantable stimulator (IS) and having the IS still in-situ (with therapy activated or deactivated) will be collected.

The main question it aims to answer is: what is the long term safety profile of the Genio System?

Participants will be asked to refer back to the site per standard of care and report on any (Serious) Adverse Device Effects and Device Deficiencies that may have occurred.

DETAILED DESCRIPTION:
The objective of this study is to assess the long-term safety of the Genio® system in adult OSA patients with and without complete concentric collapse of the soft palate who have successfully been implanted with the Genio IS in a Nyxoah sponsored Clinical Investigation.

All subjects that have previously participated in a Nyxoah sponsored clinical investigation in Australia, and who are currently still implanted with an implantable stimulator (with therapy activated or de-activated) will be asked to participate in this long-term safety follow-up study and will be asked to report any (Serious) Adverse Device Effects and Device Deficiencies that may have occurred.

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily signed an Informed Consent Form
* Subject is currently implanted with a Genio® Implantable Stimulator (IS), with therapy active or inactive, and was included in and subsequently exited a Nyxoah sponsored clinical investigation (either by study completion or withdrawal). These studies include, but are not limited to BLAST OSA (CL-GEN-001203), BETTER SLEEP (CL-GEN-001908), DREAM (CL-GEN-002033) or, subject is currently implanted with a Genio® Implantable Stimulator (IS) and accessing therapy via the TGA special access scheme (SAS).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult OSA patients with and without complete concentric collapse of the soft palate who have successfully been implanted with the Genio IS in a Nyxoah sponsored Clinical Investigation in Australia.
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-07-17 (Estimated); Study Completion 2029-07-17 (Estimated)

PRIMARY OUTCOMES:
Long-term safety | Yearly (until commercial availability of the device in Australia OR until no subjects remain implanted), anticipated average 5 years"
  Long term safety of the Genio System as measured by the rate and type of Adverse Device Effects, Serious Adverse device Effects and Device Deficiencies overtime in subjects in Australia previously implanted with a Nyxoah Genio implantable stimulator (IS) and having the IS still in-situ (with therapy activated or deactivated).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lewis, MBBS, Principal Investigator — Perth Head & Neck Surgery
Locations (7):
- Australia (7):
  - The Woolcock Institute Of Medical Research, Sydney, New South Wales
  - Westmead Public Hospital, Sydney, New South Wales
  - Illawarra ENT and Head & Neck Clinic, Sydney, New South Wales
  - Complete ENT, Brisbane, Queensland
  - Institute for Breathing and Sleep (IBAS), Melbourne, Victoria
  - Monash Health - Department of Respiratory and Sleep Medicine, Melbourne, Victoria
  - Perth Head & Neck Surgery, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No